CLINICAL TRIAL: NCT02097498
Title: Improving Patient Safety Through Simulation Research: Airway Management Proficiency Study
Brief Title: Improving Patient Safety Through Simulation Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Thomas E. Terndrup, Chair, Department of Emergency Medicine, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2013H0226
Record Dates: First submitted 2014-02-18; First posted 2014-03-27 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Airway Management Assessment
Keywords: Simulation; Enhance; Safety; Proficiency; Paramedics.; Airway Management; Intubation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Simulation only (No Intervention): One group will be randomized to receive simulation training similar to that required for certification. Paramedics in this group will then complete a second simulation scenario
- Directed feedback (Experimental): One group will review their baseline simulation scenario with a member of the research staff while providing specific feedback for errors made during the first simulation. Paramedics in this group will then complete a second simulation scenario.
  Interventions: Other: Directed feedback
- Basic Videolaryngoscopy (Experimental): One group will review a series of instructional videos related to common airway management errors. Paramedics in this group will then complete a second simulation scenario.
  Interventions: Other: Basic Videolaryngoscopy Videos

INTERVENTIONS:
Other: Directed feedback — Group will receive feedback from an airway management expert while the paramedic review their baseline simulation scenario through recorded video
  Arms: Directed feedback
Other: Basic Videolaryngoscopy Videos — Group will watch a series of educational videos related to common airway management errors.
  Arms: Basic Videolaryngoscopy

SUMMARY:
The overall objective of the present proposal is to assess whether medical simulation can enhance the safety and proficiency profile of paramedics performing prehospital endotracheal intubation, and whether feedback from an airway management expert observing the simulation enhances skill retention after 12 and 24 months. Since no validated proficiency assessment tool currently exists to measure the skill of paramedics in airway management, one will be developed and tested. Using this tool, 250 paramedics in central Ohio, will undergo simulation training similar to that required for certification. A baseline assessment of proficiency will be obtained. One group will be randomized to receive simulation training similar to that required for certification, while the other group will receive feedback from an airway management expert linked to the simulation test site via a 2-way audio-video feed. Both groups of paramedics will be reassessed at 12, and 24 months to determine whether skill level was maintained or whether skills deteriorated, and whether expert intervention had any impact on skill retention.

ELIGIBILITY:
Inclusion Criteria:

* Currently certified central Ohio paramedics

Exclusion Criteria:

* Refusal to participate
* Non-certified paramedics

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Development and validation of an airway management assessment tool | 3 years
  Employing a team of psychometric, human factors, and airway management experts, we propose to make refinements to our assessment tool so that it has objective measurement criteria, takes timing and sequencing of actions into account, provides reproducible scores, has high inter-rater reliability, and can be a valid measure of paramedic airway management proficiency and safety.

SECONDARY OUTCOMES:
Development of educational interventions to improve skill retention | 2 years
  The paramedics will be reassessed at 12 to determine whether skill level was maintained.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Terndrup, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States